CLINICAL TRIAL: NCT01992861
Title: MRI- and PET-Predictive-Assay of Treatment Outcome in Cancer of the Cervix
Brief Title: MRI and PET Imaging in Predicting Treatment Response in Patients With Stage IB-IVA Cervical Cancer
Status: Terminated | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 8118; NCI-2013-01935 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8118 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA155454 (NIH); RG3114003 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-11-05; First posted 2013-11-25 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Cervical Undifferentiated Carcinoma; Recurrent Cervical Carcinoma; Stage IB2 Cervical Cancer; Stage II Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IIIA Cervical Cancer; Stage IIIB Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic (DCE MRI, DW MRI, MR spectroscopy, FDG PET/CT): Patients undergo radiation therapy and receive chemotherapy per standard of care. Patients undergo DCE MRI, DW MRI, and MR spectroscopy at baseline, 2-2.5 weeks, 4-5 weeks, and 1 month following radiation therapy completion, and FDG PET/CT at baseline, 2-2.5 weeks, and 4-5 weeks.
  Interventions: Procedure: Computed Tomography; Procedure: Diffusion Weighted Imaging; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Radiation: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Diffusion Weighted Imaging — Undergo DW MRI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Radiation: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MR spectroscopy
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies magnetic resonance imaging (MRI) and positron emission tomography (PET) imaging in predictive treatment response in patients with stage IB-IVA cervical cancer. MRI is a procedure in which radio waves and a powerful magnet linked to a computer are used to create detailed pictures of areas inside the body. PET is a procedure in which a small amount of radioactive glucose (sugar) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is taken up. Comparing results of diagnostic procedures, such as MRI and PET, done before, during and after radiation and chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo radiation therapy and receive chemotherapy per standard of care. Patients undergo dynamic contrast-enhanced (DCE) MRI, diffusion-weighted (DW) MRI, and magnetic resonance (MR) spectroscopy at baseline, 2-2.5 weeks, 4-5 weeks, and 1 month following radiation therapy completion, and fludeoxyglucose F 18 (FDG) PET/computed tomography (CT) at baseline, 2-2.5 weeks, and 4-5 weeks.

After completion of study, patients are followed up at least every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed stage IB2-IVA epithelial carcinoma of the cervix, including squamous cell, adeno-, and undifferentiated carcinoma, and excluding small cell/neuroendocrine carcinoma, who will undergo radiation therapy for cervical cancer with curative intent
* Surgical staging with retroperitoneal staging and lymphadenectomy is permitted
* Patients who will undergo standard radiation therapy with concurrent cisplatin-based chemotherapy for cervical cancer
* Patients with no prior radiation therapy to the pelvis
* Patients with no contra-indications to magnetic resonance (MR) imaging
* Patients must have adequate renal function: glomerular filtration rate (GFR) > 30 mL/min/1.73 m^2; for the test-retest sub-study MRI, patients must have a GFR of > 60 mL/min/1.73m^2
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with small cell/neuroendocrine cervical carcinoma
* Patients who have received any prior pelvic radiation therapy in the area of the tumor that precludes the delivery of a curative dose of pelvic radiation
* Medical contraindication to MR imaging (e.g. pacemakers, metallic implants, aneurysm clips, known contrast allergy to gadolinium contrast, pregnancy, nursing mothers, weight greater than 350 pounds, GFR < 30)
* Major medical or psychiatric illness that, in the investigator's opinion, would prevent completion of treatment, completion of the study protocol, or interfere with follow-up
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IB2-IVA epithelial carcinoma of the cervix, including squamous cell, adeno-, and undifferentiated carcinoma, who will undergo radiation therapy for cervical cancer with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-02-14; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Up to 5 years
Distant metastatic rate | Up to 5 years
Local control | Up to 5 years
  Clinical/pelvic examination, pap smear, other standard of care investigations as indicated by clinical findings.
Predictive power of the MRI and PET/CT parameters | Up to 5 years
  Hazard ratios will be calculated. Predictive power of the heterogeneity metrics will be compared and ranked with Federation of Gynecology and Obstetrics stage, lymph node status, histology, hemoglobin level, and tumor anatomic volumes. Multivariate predictive algorithms will be derived by synergizing the predictive power of imaging metrics and clinical prognosticators for clinical translation.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lo, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (4):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada
- University of Hong Kong, Hong Kong, Hong Kong